CLINICAL TRIAL: NCT06089850
Title: Psychological Impact of Haploidentical Allogeneic Hematopoietic Stem Cell Transplantation on Donors
Acronym: HAPLOGREF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP211342
Record Dates: First submitted 2022-12-07; First posted 2023-10-18 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Haplo-identical Transplantation; Transplantation
Keywords: HSC transplantation; anxiety; depression; donors; hematology; familly; psychic state
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HSC donors (Experimental): Completion of questionnaires + socio-demographic data
  Interventions: Other: Evaluate the evolution of the psychic state of the donors (ascendants and descendants), by means of questionnaires, within the framework of haplo-identical allograft.

INTERVENTIONS:
Other: Evaluate the evolution of the psychic state of the donors (ascendants and descendants), by means of questionnaires, within the framework of haplo-identical allograft. — Donors are included in the study during the pre-donation assessment. Completion of questionnaires + socio-demographic data
  CSH collection visit (V1): Visit at which donors are collected for CSH donation. Completion by the donor of the questionnaires
  Follow-up of donors at D90 (+/-7) post V1, D180 (+/-15D) post V1 and D360 (+/-15D) post V1. The donors participating in the study will complete the scales/questionnaires
  D360: Completion by the donor of the questionnaires + semi-structured interview by telephone if accepted by the participant

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSC) is currently one of the only curative treatments for haematological malignancies with a poor prognosis, the realization of which presupposes the identification and availability of a compatible donor. In recent years, haploidentical transplants have been developed, a reliable alternative for patients who do not have 100% compatible donors.

The development of haplo-identical transplants leads to an exponential increase in the use of intra-family donation. Intrafamilial donation of hematopoietic stem cells (HSC) has the advantages of lower financial cost and faster availability of the graft, thus avoiding the risk of relapse before the procedure. Nevertheless, intrafamilial donation raises clinical and ethical questions. Indeed, the psychological impact of intra-family donation on the donor cannot be overlooked. Thus, in the context of the development of haplo-identical transplants, measuring the impact of donation on donors (ascendants and descendants) will make it possible to assess the relevance of taking psychosocial aspects into consideration in the choice of donors, to assess the psychological impact of haplo-identical donation and to offer psychological support adapted to donors.

DETAILED DESCRIPTION:
This is a prospective, exploratory and bicentric study with a quantitative and qualitative approach, with the aim of exploring the psychosocial aspects of the experience of haplo-identical transplantation in adult HSC donors for transplantation. haplo-identical for their children or for their parents.

For this, the evolution of the anxiety and depression) of the donors will be evaluated on D0, D90, D180 and D360 post donation, thanks to State-Trait anxiety Inventory questionnaire, Center for Epidemiologic Studies Depression Scale and by the 12-Item Short Form Health Survey;

ELIGIBILITY:
Inclusion criteria:

* Identical haplo CSH donors ascending (parents) or descending (children)
* Major identical haplo HSC donors
* Haplo-identical HSC donors living in mainland France and cared for in the centers participating in the study
* Haplo-identical HSC donors benefiting from Social Security System.
* Haplo-identical HSC donors who have signed the consent form
* - Ability to read and write in French

Exclusion Criteria:

- Insufficient understanding of the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety | D0 ; D90, D180 and D360
  Assessed by the State-Trait anxiety Inventory (STAI-Y), self-questionnaire validated in French
  STAI-Y : Spielberger trait anxiety questionnaire minimum value : almost never maximum value : almost always Higher score = better outcome

SECONDARY OUTCOMES:
Depression | Day 360
  Assessed by the Center for Epidemiologic Studies Depression Scale (CES-D self-questionnaire) validated in French
  CES-D : Center for Epidemiologic Studies -Despression Minimum value : never (0) Maximum value : all the time (3)
  Coding (except questions 4/8/12/16):
  * Never = 0 pts
  * Very rarely (less than 1 day) = 0 pts
  * Occasionally (1 to 2 days) = 1 pts
  * Quite often (3 to 4 days) = 2 pts
  * Frequently (5 to 7 days) = 3 pts
  * All the time = 3 pts
  Coding questions 4/8/12/16:
  * Never = 3 pts
  * Very rarely (less than 1 day) = 3 pts
  * Occasionally (1 to 2 days) = 2 pts
  * Quite often (3 to 4 days) = 1 pts
  * Frequently (5 to 7 days) = 0 pts
  * Constantly = 0 pts
  Higher score = worse outcome
Quality of donor's life | Day 360
  Assessed by the 12-Item Short Form Health Survey (SF-12), validated for the French population SF-12 : quality of life It is a quality of life questionnaire and no score is reported on a scale
Family functioning | Day 360
  Explored by semi-structured telephone interview
Describe the donor management methods | Day 0
  Sheet to be completed by the participating centers
Describe the symptoms experienced during the administration of the growth factor and the collection of HSCs | Day 90
  Questionnaire to be completed by the donors
Describe the medical problems encountered since the donation of HSCs | Day 360
  Questionnaire to be completed by donors
Evaluate the donors' perception of the care offered to them | Day 360
  Questionnaire to be completed by donors
  FRI : French adaptation of the Family Relationship Index Scale : true (1)/False (0) A high score indicates respectively: high family cohesion, high expression/verbalization of feelings, high conflict and good family relationships.
  * Describe the donor management methods : no scale
  * Describe the symptoms experienced during the administration of the growth factor and the collection of HSCs (questionnaire B at D90) : no scale. It is a questionnaire where the donor describes his feelings during the administration of the growth factor
  * Describe the medical problems encountered since the donation of HSC (questionnaire C at D180 and 360) : no scale, It is a questionnaire in which the donor describes any medical problems encountered since the donation
  * Evaluate the donors' perception of the care offered to them (questionnaire D at D360) : no scale, This is a questionnaire that the patient answers in order to improve donor management.
Describe the medical events concerning the donation of CSH | Day 360
  Questionnaire to be completed by donors
Describe medical events in patients and assess the impact on the donor's mental state | Day 360
  Collect information on the patient journey (GVH, relapse, death)
  The experiences of the donors will be explored through semi-structured interviews, the interest of the qualitative approach having been demonstrated for an in-depth understanding of the psychological problems.

CONTACTS AND LOCATIONS:
Overall Officials: Eolia Brissot, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service D'hématologie Clinique et thérapie cellulaire - Hôpital St Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided